CLINICAL TRIAL: NCT07247422
Title: Cardioneural Temporary Pacing to Achieve Autonomic Modulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tam Tsz Kin, Prof, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Temp CNP Study
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Temporary Cardio-neural Pacing; Pacemaker Implantation
Keywords: cardio-neural pacing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- temporary cardio-neural pacing (Experimental): Patient will undergo temporary cardio-neural pacing in study procedure
  Interventions: Procedure: Temporary cardio-neural pacing

INTERVENTIONS:
Procedure: Temporary cardio-neural pacing — Arterial line will be inserted for monitoring of blood pressure. A temporary ventricular lead will be first implanted, potentially to the left bundle area to preserve normal conduction physiology. A coronary sinus sheath (attain command or deflectable) will be delivered to RA septum, posterior to CS ostium, at the expected location of parasympathetic ganglion plexus. Pace mapping will be performed with a pacing lead (such as Select Secure 3830) at 30Hz. An electrophysiology catheter may be used where necessary for pace-mapping the response. At the site where lowest output can generate 30% prolongation of ventricular CL, the lead is fixed for 1-5mm depth. The output is tested again to achieve heart rate slowing to less than 80bpm. Fluoroscopic image will be collected with contrast injection at the sheath. Eventually, the implanted lead will be connected into a temporary pacemaker. The temporary leads will be removed when no longer clinically required.

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia, with a lifetime risk of 1 in 3-5. In cases of rapid ventricular rate, patients often experience low blood pressure, making standard rate and rhythm control medications contraindicated. While cardioversion may be necessary, it is often ineffective in long-standing AF and can lead to left ventricular stunning. This creates a vicious cycle, worsening heart failure and cardiogenic shock.

AV node ablation may be required, but it is irreversible and carries risks, including complications from long-term pacing. Therefore, temporary pacing may be a preferable option to allow for hemodynamic improvement and better ventricular filling.

Research suggests that parasympathetic fibers innervating the AV node can modulate conduction. Ablation in these fibers has shown promise for treating vagal-mediated syncope, and high-frequency pacing may provide chronic heart rate suppression. Intermittent pacing has also been effective in reducing ventricular rates in atrial fibrillation to prevent inappropriate ICD shock. This may be potentially beneficial for patients with uncontrolled fast AF.

In a proof-of-concept study with five patients, pacing at 30Hz and 10mA in the coronary sinus resulted in a dose-dependent prolongation of the ventricular cycle length during AF, with stable blood pressure and no discomfort reported. This suggests that pacing these fibers could achieve rate control without the need for medications or AV node ablation, with no complications observed.

This study aims to evaluate safety and efficacy of temporary cardio-neural pacing (CNP). This is a prospective cohort study involving patients with atrial fibrillation (AF) and rapid ventricular conduction who have failed or are contraindicated for rate control with antiarrhythmic medications. Enrolled patients will be followed up for 1 month.

DETAILED DESCRIPTION:
During procedure, arterial line will be inserted for monitoring of blood pressure. A temporary ventricular lead will be first implanted, potentially to the left bundle area to preserve normal conduction physiology. A coronary sinus sheath (attain command or deflectable) will be delivered to RA septum, posterior to CS ostium, at the expected location of parasympathetic ganglion plexus. Pace mapping will be performed with a pacing lead (such as Select Secure 3830) at 30Hz. An electrophysiology catheter may be used where necessary for pace-mapping the response. At the site where lowest output can generate 30% prolongation of ventricular CL, the lead is fixed for 1-5mm depth. The output is tested again to achieve heart rate slowing to less than 80bpm. Fluoroscopic image will be collected with contrast injection at the sheath. Eventually, the implanted lead will be connected into a temporary pacemaker. The temporary leads will be removed when no longer clinically required, such as when the heart rate stabilized. Cardioneural pacing will be performed at lowest output at a frequency of 5-50Hz via the atrial lead (CNP lead). The ventricular lead will have pacing mode being set at 80bpm VVI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrial fibrillation or atrial flutter who are having rapid ventricular rate >100bpm
* Patient who cannot take rate control agents, or heart rate control remains unsatisfactory after rate control agents

Exclusion Criteria:

* Patients who cannot provide informed consent
* Patients < 18 years old
* Pregnant patients
* Illiterate patients

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Heart Rate equal or lower than 80bpm | In implant procedure
  Number of patients achieving <=80bpm heart rate with cardio-neural pacing

SECONDARY OUTCOMES:
Threshold | In implant procedure
  Pacing threshold to achieve HR<=80 with CNP.
Patient discomfort | In implant procedure
  Number of patients with discomfort from patient during CNP
Mean blood pressure | In implant procedure
  Mean blood pressure during CNP, compared with that before pacing.
Blood Biochemistry | In implant procedure
  Change of blood biochemistry including lactate level and pH in blood gas.
Inotrope dosage | In implant procedure
  Determine Inotrope dosage

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Sha Tin, Hong Kong